CLINICAL TRIAL: NCT02581462
Title: FLOT vs. FLOT/Herceptin/Pertuzumab for Perioperative Therapy of Adenocarcinoma of the Stomach and Gastroesophageal Junction Expressing HER-2. A Phase II/III Trial of the AIO.
Brief Title: FLOT vs. FLOT/Herceptin/Pertuzumab for Perioperative Therapy of HER-2 Expressing Gastric or GEJ Cancer
Acronym: PETRARCA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Collaborators: Trium Analysis Online GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML29452/PETRARCA/FLOT6
Record Dates: First submitted 2015-10-19; First posted 2015-10-21 (Estimated); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Stomach Cancer; Gastroesophageal Junction Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Trastuzumab; pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FLOT alone (Experimental): Pre-operative therapy with FLOT followed by surgical resection followed by post-operative therapy with FLOT
  Interventions: Drug: FLOT alone
- FLOT + Herceptin/Pertuzumab (Experimental): Pre-operative therapy with FLOT + Herceptin/Pertuzumab followed by surgical resection followed by post-operative therapy with FLOT + Herceptin/Pertuzumab
  Interventions: Biological: FLOT + Herceptin/Pertuzumab

INTERVENTIONS:
Drug: FLOT alone — Pre-operative therapy:
  * Docetaxel 50 mg/m², d1, d15, d29, d43
  * Oxaliplatin 85 mg/m², d1, d15, d29, d43
  * Leucovorin 200 mg/m², d1, d15, d29, d43 (can be replaced by sodium folinate according to local guidelines)
  * 5-FU 2600 mg/m², d1, d15, d29, d43
  Surgery is recommended to be scheduled 4 weeks after d43.
  Post-operative therapy (start 6 to 8 weeks after surgery):
  * Docetaxel 50 mg/m², d1, d15, d29, d43
  * Oxaliplatin 85 mg/m², d1, d15, d29, d43
  * Leucovorin 200 mg/m², d1, d15, d29, d43 (can be replaced by sodium folinate according to local guidelines)
  * 5-FU 2600 mg/m², d1, d15, d29, d43
  Arms: FLOT alone
Biological: FLOT + Herceptin/Pertuzumab — Pre-operative therapy:
  * Herceptin 8/6 mg/kg, d1, d22, d43
  * Pertuzumab 840 mg, d1, d22, d43
  * Docetaxel 50 mg/m², d1, d15, d29, d43
  * Oxaliplatin 85 mg/m², d1, d15, d29, d43
  * Leucovorin 200 mg/m², d1, d15, d29, d43 (can be replaced by sodium folinate according to local guidelines)
  * 5-FU 2600 mg/m², d1, d15, d29, d43
  Surgery is recommended to be scheduled 4 weeks after d43.
  Post-operative therapy (start 6 to 8 weeks after surgery):
  * Herceptin 8/6 mg/kg, d1, d22, d43
  * Pertuzumab 840 mg, d1, d22, d43
  * Docetaxel 50 mg/m², d1, d15, d29, d43
  * Oxaliplatin 85 mg/m², d1, d15, d29, d43
  * Leucovorin 200 mg/m², d1, d15, d29, d43 (can be replaced by sodium folinate according to local guidelines)
  * 5-FU 2600 mg/m², d1, d15, d29, d43.
  Arms: FLOT + Herceptin/Pertuzumab

SUMMARY:
Previous studies provide a strong theoretical rationale for the conduct of a randomized study evaluating the efficacy and safety of Herceptin and pertuzumab in combination with FLOT in the perioperative treatment of resectable HER-2 positive adenocarcinoma of the stomach or GEJ.

DETAILED DESCRIPTION:
This is a multicenter, randomized, controlled, open-label study including patients with locally advanced adenocarcinoma of the stomach and GEJ scheduled to receive perioperative chemotherapy. According to centrally assessed HER-2 status: Patients with HER-2 positive tumors will receive FLOT +/- Herceptin / pertuzumab.

The scope of the phase II portion of the trial is to evaluate pathological response rates of either regimen assessed by a centralized pathology and define safety and tolerability.

Patients with locally advanced esophagogastric adenocarcinoma (i.e. cT2 any N or any T N-positive) with exclusion of distant metastases will be included in this trial.

Patients will be stratified by age (18-69 vs. ≥ 70), tumor site (GEJ vs. gastric) and clinical stage (T1/2 vs. 3/4 and N- vs. N+) and randomized 1:1 to receive either FLOT (Arm A) or FLOT/Herceptin/pertuzumab (Arm B).

Arm A (control group) Patients randomized to Arm A will receive 4 pre-operative treatments of FLOT (Docetaxel 50 mg/m², iv over 2 h; Oxaliplatin 85 mg/m² in 500 ml G5%, iv over 2h; Leucovorin 200 mg/m² in 250 ml NaCl 0.9 %, iv over 1 h; 5-FU 2600 mg/m², iv over 24 h) on d1, d15, d29, d43 of the preoperative treatment phase. Surgery is recommended to occur 4 weeks after last FLOT (4 weeks after d43 = day 71). Patients will receive 4 additional post-operative treatments of FLOT on d1, d15, d29, and d43 of the post-operative treatment phase. Post-operative treatment should start 6 to 8 weeks, but at maximum 12 weeks after surgery.

Arm B (Herceptin/pertuzumab group) Patients randomized to Arm B will receive the FLOT regimen identical to Arm A as described above in conjunction with three-weekly Herceptin at 8mg/kg initial dose (Day 1, loading dose) followed by subsequent doses of Herceptin at 6mg/kg on d22 and d43 and pertuzumab at 840mg on d1, d22, and d43. Surgery is recommended to occur 4 weeks after last FLOT/Herceptin/pertuzumab dose (4 weeks after d43 = day 71). Patients will receive 3 additional doses of Herceptin and pertuzumab on d1, d22, and d43 of the post-operative treatment phase, together with the postoperative chemotherapy. Moreover, patients will receive 11 additional doses of Herceptin and pertuzumab after the end of post-operative FLOT.

In both of the arms, tumor assessments (CT or MRI) are performed before randomization and prior to surgery and then every 3 months thereafter until progression/relapse, death or end of follow-up.

During treatment, clinical visits (blood cell counts, detection of toxicity) occur prior to every treatment dose. Safety of FLOT/Herceptin/pertuzumab will be monitored continuously by careful monitoring of all adverse events (AEs) and serious adverse events (SAEs) reported.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the GEJ (type I-III) or the stomach (uT2, uT3, uT4, any N category, M0), or any T N+ M0 patient, with the following specifications:

   * Medical and technical operability
   * Centralized detection of either an adenocarcinoma with HER-2 3+ (IHC) or HER-2 2+ (IHC) with amplification proven by FISH, SISH or CISH
2. No preceding cytotoxic or targeted therapy
3. No prior partial or complete tumor resection
4. Exclusion of the infiltration of any adjacent organs or structures by CT or MRI
5. Exclusion of distant metastasis by CT or MRI of thorax and abdomen, and bone scan (if osseous lesions are suspected due to clinical signs)
6. Female and male patients ≥ 18 years. Patients in reproductive age must be willing to use adequate contraception during the study and for 7 months after the end of pertuzumab and Herceptin treatment (Appropriate contraception is defined as surgical sterilization (e.g., bilateral tubal ligation, vasectomy), hormonal contraception (implantable, patch, oral), and double-barrier methods (any double combination of: IUD, male or female condom with spermicidal gel, diaphragm, sponge, cervical cap)). Female patients with childbearing potential need to have a negative pregnancy test within 7 days before study start.
7. ECOG ≤ 2
8. Laparoscopic exclusion of peritoneal carcinomatosis, if suspected clinically
9. Adequate haematological, hepatic and renal function parameters:

   * Leukocytes ≥ 3.000/mm³, platelets ≥ 100.000/mm3
   * Serum creatinine ≤ 1.5 x upper limit of normal, or GFR > 40 ml/min
   * Bilirubin ≤ 1.5 x upper limit of normal, AST and ALT ≤ 3.5 x upper limit of normal, alkaline phosphatase ≤ 6 x upper limit of normal
10. LVEF value > 55 %, as assessed by echocardiography
11. Patient able and willing to provide written informed consent and to comply with the study protocol and with the planned surgical procedures

Exclusion Criteria:

1. Patients with involved retroperitoneal (e.g. para-aortal, paracaval or interaortocaval lymph nodes) or mesenterial lymph nodes (distant metastasis!)
2. Known hypersensitivity against Herceptin, pertuzumab, 5-FU, leucovorin, oxaliplatin, or docetaxel
3. Other known contraindications against Herceptin, pertuzumab, 5-FU, leucovorin, oxaliplatin, or docetaxel
4. Documented history of congestive heart failure of any NYHA, myocardial infarction within the past 6 months before the first dose of study treatment
5. Clinically significant valvular defect , history of poorly controlled arterial hypertension (systolic blood pressure > 180 mmHG or diastolic blood pressure > 100 mmHg) or uncontrollable high-risk cardiac arrhythmia (i.e tachycardia with a heart rate > 100/min at rest), significant ventricular arrhythmia (ventricular tachycardia) or higher grade atrioventricular-block (second degree AV-block Type 2 (Mobitz2) or third degree AV-block)
6. Past or current history of other malignancies not curatively treated and without evidence of disease for more than 5 years, except for curatively treated basal cell carcinoma of the skin and in situ carcinoma of the cervix
7. Known brain metastases
8. Other severe internal disease or acute infection
9. Peripheral polyneuropathy ≥ NCI Grade II
10. Chronic inflammatory bowel disease
11. Clinically significant active GI bleeding
12. On-treatment participation in another clinical study in the period 30 days prior to inclusion and during the study
13. Subject pregnant or breast feeding, or planning to become pregnant within 6 months after the end of treatment.
14. Patients in a closed institution according to an authority or court decision (AMG § 40, Abs. 1 No. 4)
15. Any other concurrent antineoplastic treatment including irradiation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2020-07-17 (Actual)

PRIMARY OUTCOMES:
PhaseII: Rate of pathological complete response | 3 years
Phase III: Median Progression Free Survival | 5 years

SECONDARY OUTCOMES:
Phase II/III: R0 resection rate | 75 days
Phase II: Median Progression Free Survival (PFS) | 3 years
Phase II/III: Median Overall Survival | 3/5 years
Phase II: PK Analysis | 3 years
Phase II/III: Subgroup analyses: pathological response according to HER-2 status HER-2 IHC 3+ vs. other cases | 3/5 years
Phase II/III: Subgroup analyses: PFS according to HER-2 status HER-2 IHC 3+ vs. other cases | 3/5 years
Phase II/III: Subgroup analyses: OS according to HER-2 status HER-2 IHC 3+ vs. other cases | 3/5 years
Phase III: Pathological Response Rates | 5 years
Phase III: PFS rates | 3 and 5 years
Phase III: OS rates | 3 and 5 years
Phase III: Median OS | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Salah-Eddin Al-Batran, Prof. Dr., Study Chair — Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest
Locations (1):
- Institute for Clinical Cancer Research Krankenhaus Nordwest, Frankfurt, Germany

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.

REFERENCES:
- [Derived] Hofheinz RD, Merx K, Haag GM, Springfeld C, Ettrich T, Borchert K, Kretzschmar A, Teschendorf C, Siegler G, Ebert MP, Goekkurt E, Mahlberg R, Homann N, Pink D, Bechstein W, Reichardt P, Flach H, Gaiser T, Battmann A, Oduncu FS, Loose M, Sookthai D, Pauligk C, Goetze TO, Al-Batran SE. FLOT Versus FLOT/Trastuzumab/Pertuzumab Perioperative Therapy of Human Epidermal Growth Factor Receptor 2-Positive Resectable Esophagogastric Adenocarcinoma: A Randomized Phase II Trial of the AIO EGA Study Group. J Clin Oncol. 2022 Nov 10;40(32):3750-3761. doi: 10.1200/JCO.22.00380. Epub 2022 Jun 16. PMID 35709415